CLINICAL TRIAL: NCT06985017
Title: Playing Playfully to Overcome Adversity
Acronym: PPOA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sacred Heart University (Other)
Collaborators: Yeshiva University (Other)
Responsible Party: Principal Investigator, Lola Halperin, Ed.D., OTR/L, Assistant Professor, Sacred Heart University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 210413A
Record Dates: First submitted 2025-05-12; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Adverse Childhood Experiences
Keywords: Childhood adversity, teacher training, play, playfulness

STUDY DESIGN:
Intervention Model Description: The training program used in this study aims to equip teachers serving children exposed to adversity with the knowledge and skills pertaining to using play and playfulness as vehicles to foster children's growth. NO DRUGS ARE INVOLVED IN THIS STUDY.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Playing Playfully to Overcome Adversity, Online Teacher Training program (Experimental): Forty five minute-long group training sessions conducted by one of the PI-s via Zoom, once a week over five weeks.
  Interventions: Behavioral: Playing Playfully to Overcome Adversity

INTERVENTIONS:
Behavioral: Playing Playfully to Overcome Adversity — This training is provided via virtual group sessions (Telehealth) and consists of five 45-minute-long weekly sessions addressing ways to promote children's play and playfulness in the classroom and techniques to reduce teacher/caregiver burnout.

SUMMARY:
This research project was developed in an effort to support teachers of young children exposed to adversity and to assist them with enhancing children's development through play. The project utilizes an occupational therapist-led teacher training program manual and an accompanying fidelity checklist. This training is provided via virtual group sessions (Telehealth) and consists of five 45-minute-long sessions addressing ways to promote children's play and playfulness in the classroom and techniques to reduce teacher/caregiver burnout. The training was facilitated via Zoom with eleven teachers employed by an agency serving children exposed to adversity. The fidelity raters scored the fidelity checklist while reviewing video recordings of the training sessions. Participants responded to a Background Questionnaire via Qualtrics and were interviewed before and after the training. The interview data was used to analyze the impact of the training.

DETAILED DESCRIPTION:
This pilot study examines the feasibility of a teacher group training program that aims to equip teachers with the skills of promoting development among young children exposed to adversity through play. The study utilizes occupational therapist-led teacher training program manual entitled Playing Playfully to Overcome Adversity (PPOA) and an accompanying fidelity checklist. This training is provided via virtual group sessions (Telehealth) and consists of five 45-minute-long sessions addressing ways to promote children's play and playfulness in the classroom.

The project's goals are:

1. To determine whether the above program can:

   1. Increase teachers' perceived competencies supporting play in the classroom
   2. Change teachers' views of how they can support children's play and playfulness
2. To identify program elements that require revisions/modifications based on teachers' feedback pertaining to:

   1. Aspects of the program that they find to be helpful or less helpful
   2. Aspects of the training they deem to be feasible to implement in their classrooms in order to promote children's play and playfulness

The PPOA training was facilitated via Zoom with eleven teachers employed by an agency serving children exposed to adversity. The fidelity checklist was scored while reviewing video recordings of the training sessions. Participants responded to a Background Questionnaire via Qualtrics and were interviewed before and after the training. Interview data was used to analyze the impact of the training.

ELIGIBILITY:
Inclusion Criteria:

* Teachers and teacher assistants employed by agencies serving young children exposed to adversity who have access to a device with reliable high-speed internet, camera, and Zoom capacity.

Exclusion Criteria:

* Individuals who are not teachers or teacher assistants employed by agencies serving young children exposed to adversity or who do not have access to a device with reliable high-speed internet, camera, and Zoom capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Parent/Caregiver's View of Supporting Children's Play and Playfulness | From enrollment to the end of treatment at 6 weeks
  The questionnaire assesses parent or caregiver perception of their support of child's playfulness. It consists of 11 items scored on 3-point scale ranging from 0 (do not agree) to 2 (strongly agree).
Teacher Perception of Play in the Classroom Survey | From enrollment to the end of treatment at 6 weeks
  The Teacher Perception of Play in the Classroom Survey assesses teachers' confidence in incorporating play and/or playful attitude into the classroom environment. It consists of 14 statements on a 3-point scale ranging from 1 (not true) to 3 (certainly true).

SECONDARY OUTCOMES:
Open-ended pre-program questions | At enrollment
  Three pre-training participant interview questions about their beliefs pertaining to play's role in children's development, what play looks like in their classroom, and what they expect to gain from participating in the training program.
Post-Training Participant Interview | After 6 weeks
  A set of seven post program questions to learn on the benefits of the program and areas for improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Amiya Waldman-Levi, PhD, Principal Investigator — Yeshiva University
Locations (1):
- Sacred Heart University, Fairfield, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be shared through publications.

REFERENCES:
- [Background] Halperin L, Waldman-Levi A. Playing Playfully to Overcome Adversity: A Telehealth-Based Group Teacher Training Program. OTJR (Thorofare N J). 2023 Jul;43(3):381-389. doi: 10.1177/15394492231151882. Epub 2023 Feb 7. PMID 36748710